CLINICAL TRIAL: NCT05823558
Title: Comparison of Lumbar Muscle Thickness Measurements in Osteoporotic and Osteopenic Patients
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aylin Ayyıldız, Medical Doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 10042023
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Ostoporotic Patients Group: T value of -2.5 and below in DEXA measurement
  Interventions: Diagnostic Test: Lomber Muscle Thickness Measurement
- Osteopenic Patients Group: T value between -2.5 and -1 in DEXA measurement
  Interventions: Diagnostic Test: Lomber Muscle Thickness Measurement
- Healthy Group: T value of -1 and above in DEXA measurement
  Interventions: Diagnostic Test: Lomber Muscle Thickness Measurement

INTERVENTIONS:
Diagnostic Test: Lomber Muscle Thickness Measurement — Muscle thickness measurements will be made on the imaging of those who have lumbar MR imaging.

SUMMARY:
In osteoporosis, sarcopenia is a common condition. Sarcopenic measurements can be made by evaluating muscle thickness in different regions. We aim to evaluate lumbar muscle losses in patients with osteoporosis in the lumbar region and to examine whether these muscle losses are correlated with the level of osteoporosis. The patients will be divided into 3 groups as healthy, osteopenic and osteoporotic according to DEXA measurements. Demographic values, comorbidities, osteoporosis drugs used, fracture histories, L1-4, L2-4, femoral neck and total BMD and t values of the patients, psoas and multifidus muscle measurements will be made at L2-L3 level in Lumbar MR imaging. Lumbar MR muscle measurements will be made by 1 physician blind to the DEXA values of the patients.

ELIGIBILITY:
Inclusion Criteria:

* 50-90 years old
* 2. Recent MRI of the lumbar region with DEXA evaluation

Exclusion Criteria:

* Have had previous lumbar surgery
* Any previous lumbar injection
* Stage 3-4 Lumbar Listesis
* Presence of Lumbar Discopathy accompanied by neurological deficit

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50-90 years old osteoporotic, osteopenic and healthy people
Sampling Method: Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Lomber Muscle Measurement | Day 1
  Psoas and multifidus muscle measurements will be made at L2-L3 level in Lumbar MR imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Etfal Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No